CLINICAL TRIAL: NCT06663345
Title: A Comparison of the Effects of TAP (Transversus Abdominis Plane) Block and QLB-1 (Lateral Quadratum Lumbarum) Block on Postoperative Pain and Opioid Consumption in Laparoscopic Cholecystectomy
Brief Title: Effects of TAP and QLB-1 Blocks on Opioid Consumption
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Başakşehir Çam & Sakura City Hospital (Other Government)
Responsible Party: Principal Investigator, Emine OZCAN, Principal Investigator, Başakşehir Çam & Sakura City Hospital
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Prevention
Other Study IDs: EK3419
Record Dates: First submitted 2024-07-01; First posted 2024-10-29 (Actual); Last update posted 2026-01-06 (Actual); Status verified 2026-01

CONDITIONS: Postoperative Pain
Keywords: TAP (transversus abdominis Plane) block; QLB-1 (Lateral Quadratum Lumborum ) block; Nonopioid analgesia; postoperative pain; laparoscopic cholecystectomy
MeSH Terms: conditions — Pain, Postoperative; Bites and Stings | interventions — 1,3-bis(4-amidinophenoxy)-2-(4-amidinophenoxymethyl)ethylpropane; Dental Occlusion

STUDY DESIGN:
Intervention Model Description: Prospective Randomized
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- TAP (Transversus Abdominis Plan) Block (Active Comparator): A bilateral TAP or QLB-1 block will be performed. This block is a standard procedure in our hospital for the management of postoperative pain.
  Interventions: Procedure: Transversus Abdominis Plan Block (TAPB), Lateral Quadratum Lumborum (QLB-1) Block
- QLB-1 (Lateral Quadratum Lumborum ) Block (Experimental): Investigation of the efficacy of QLB-1 block compared to TAP block.
  Interventions: Procedure: Transversus Abdominis Plan Block (TAPB), Lateral Quadratum Lumborum (QLB-1) Block

INTERVENTIONS:
Procedure: Transversus Abdominis Plan Block (TAPB), Lateral Quadratum Lumborum (QLB-1) Block — Following the acquisition of informed consent prior to surgery, 2 mg of intravenous midazolam will be administered to patients who volunteer. These patients will be monitored in the preoperative preparation room. Bilateral TAP or QLB-1 block will be performed, and this block is routinely applied for postoperative pain in our hospital.

SUMMARY:
Laparoscopic cholecystectomy is associated with less pain than open surgery and a shorter recovery time. While the type of pain experienced after laparoscopy differs from that experienced after laparotomy, it is predominantly parietal pain (originating from the abdominal wall). However, patients also report visceral pain due to pneumoperitoneum. Various analgesic procedures, including nonsteroidal anti-inflammatory drugs (NSAIDs), opioids, and regional anesthesia techniques, are employed as part of multimodal analgesia for postoperative pain. Regional anesthesia techniques for abdominal surgery include thoracic epidural analgesia, paravertebral block, and transversus abdominis plane (TAP) block. TAP block, one of the truncal blocks, has been utilized in numerous studies in the literature for the management of postoperative pain following abdominal surgery. TAPB is a nerve block technique that blocks sensory nerves by injecting local anesthetic into the plane between the transverse abdominis and internal oblique muscles. Although TAPB can effectively relieve somatic pain in patients undergoing minimally invasive laparoscopic surgery, it may not be suitable for visceral analgesia. Another truncal block that has gained recent attention is the Quadratus Lumborum Block (QLB). QLB is another nerve block technique that blocks sensory nerves by injecting local anesthetic into the interfascial plane between the quadratus lumborum and psoas muscles. QLB offers several advantages, including the ability to provide both somatic and visceral analgesia. This comprehensive approach can result in more effective postoperative analgesia during laparoscopic surgical procedures. Additionally, the use of TAPB or QLB may reduce opioid consumption, potentially improving analgesia in laparoscopic surgeries. The quadratus lumborum muscle can be blocked in four different ways: lateral, posterior, anterior, and intramuscular. In our study, the lateral quadratus lumborum block was the preferred approach. Opioids are the most commonly used narcotic analgesics for postoperative pain. Patients often require opioids for pain relief in the perioperative period, especially in abdominal surgery. However, the use of opioids can lead to a variety of side effects, including excessive sedation, postoperative nausea and vomiting, urinary retention, constipation, hyperalgesia, respiratory depression and immunosuppression. Opioids may have various effects on immune function, including modulation of cytokines, interaction with immune cells, affecting the neuroendocrine system and vascular permeability. These effects may contribute to postoperative complications such as infections and delayed wound healing due to increased inflammatory response. They may also prolong hospitalization. In order to reduce postoperative opioid consumption and opioid-related side effects, ultrasound-guided trunk block techniques are being developed in abdominal surgeries. Currently, ultrasound-guided multimodal analgesia techniques are widely used. Transversus abdominis plane block (TAPB) and quadratus lumborum block (QLB) are effective analgesic methods employed in conjunction with multimodal analgesia techniques during anesthesia. The objective of this study was to compare the effects of TAPB (transversus abdominis plane block) and QLB-1 (lateral quadratus lumborum block), which are frequently used in our clinic, on postoperative pain scores and the need for additional analgesics. Secondary objectives included postoperative opioid consumption, nausea and vomiting, hospital stay, and patient and surgeon satisfaction.

ELIGIBILITY:
Inclusion Criteria:

* - Consenting patients,
* He's having a laparoscopic cholecystectomy,
* ASA-I-II,
* Between the ages of 18 and 64,
* No history of anticoagulant or antiaggregant drug use,
* Regional anesthesia is not contraindicated and the anesthesiologist is deemed appropriate for regional anesthesia,
* Under general anesthesia and undergoing laparoscopic surgery,
* Oriented and cooperative patients,

Exclusion Criteria:

* - Patients without consent
* Regional anesthesia is contraindicated,
* He's having open abdominal surgery,
* Not in the appropriate age range,
* Chronic diseases such as uncontrolled DM and HT,
* Drug allergy,
* Taking anticoagulants or antiaggregants,
* History of chronic analgesic use,
* Presence of active infection in the area to be blocked,
* Will not be able to comply with postoperative pain /VAS follow-up,
* Patients with ASA-IV-V

Ages: 18 Years to 64 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 60 (Estimated)
Dates: Start 2024-12-25 (Actual); Primary Completion 2026-03-25 (Estimated); Study Completion 2026-07-28 (Estimated)

PRIMARY OUTCOMES:
A comparison of the effects of TAP (Transversus Abdominis Plane) block and QLB-1 (Lateral Quadratum Lumbarum) block and opioid consumption in laparoscopic cholecystectomy. | 02.11.2024 - 02.05.2025 ( 6 months)
  Rate of opioid analgesic use mg/kg/day
A comparison of the effects of TAP (Transversus Abdominis Plane) block and QLB-1 (Lateral Quadratum Lumbarum) block on postoperative pain in laparoscopic cholecystectomy. | 02.11.2024 - 02.05.2025 ( 6 months)
  Pain Measures VAS (Visual Analog Scale) Minimum: 0- Maximum: 10

CONTACTS AND LOCATIONS:
Overall Officials: Emine OZCAN, Principal Investigator — Başakşehir Çam & Sakura City Hospital
Locations (1):
- Başakşehir Çam ve Sakura Şehir Hastanesi, Istanbul, Başakşehir, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Gao T, Wang Y, Zheng Y, Yu Y, Li Q, Zhang L. Quadratus lumborum block vs. transversus abdominis plane block for postoperative pain control in patients with nephrectomy: A systematic review and network meta-analysis. J Clin Anesth. 2024 Aug;95:111453. doi: 10.1016/j.jclinane.2024.111453. Epub 2024 Mar 25. PMID 38531283
- [Background] Marcolin P, Amaral S, Motter SB, Brandao GR, de Oliveira Trindade B, Messer N, Poli de Figueiredo SM. Quadratus lumborum block versus transversus abdominis plane block for inguinal hernia repair: A systematic review and meta-analysis with trial sequential analysis. World J Surg. 2024 Mar;48(3):610-621. doi: 10.1002/wjs.12064. Epub 2024 Jan 24. PMID 38265244
- [Background] Dai J, Lin S, Cui X, Xu Z, Zheng R, Wu D. The effects of ultrasound-guided QLB and TAPB combined with opioid-free anesthesia (OFA) on clinical efficacy of the patients undergoing abdominal surgery. Heliyon. 2023 Oct 11;9(10):e20878. doi: 10.1016/j.heliyon.2023.e20878. eCollection 2023 Oct. PMID 37867884
- [Background] Sertcakacilar G, Yildiz GO. Analgesic efficacy of ultrasound-guided transversus abdominis plane block and lateral approach quadratus lumborum block after laparoscopic appendectomy: A randomized controlled trial. Ann Med Surg (Lond). 2022 Jun 14;79:104002. doi: 10.1016/j.amsu.2022.104002. eCollection 2022 Jul. PMID 35860161

DOCUMENTS (1):
  • Informed Consent Form (2024-06-06): https://cdn.clinicaltrials.gov/large-docs/45/NCT06663345/ICF_000.pdf